CLINICAL TRIAL: NCT02016495
Title: Efficacy of Magnesium and Alpha Lipoic Acid Supplementation in Reducing Premature Uterine Contractions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Responsible Party: Sponsor
Other Study IDs: Mg-ALA
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-10

CONDITIONS: Pregnancy
MeSH Terms: interventions — Magnesium; Thioctic Acid

ARMS (2):
- Magnesium + Lipoic Acid (Active Comparator)
  Interventions: Dietary Supplement: Magnesium plus alpha-lipoic acid
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium plus alpha-lipoic acid
  Arms: Magnesium + Lipoic Acid
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate whether a combined supplementation of magnesium and lipoic acid is able to significantly reduce the incidence of uterine contractions and related episodes of hospitalization in pregnant women.

DETAILED DESCRIPTION:
Primary prevention of preterm labor is based on the early identification of risk factors and on appropriate treatments. Although several drugs are currently used, the identification of effective and safe agents able to improve both maternal and fetal health is still warranted.

In this study the efficacy a formulation based on magnesium and alpha-lipoic acid has been compared with placebo to evaluate the incidence of reduction of preterm delivery.

Three hundred pregnant women at 14-34 weeks of gestation were enrolled and randomly divided to receive a daily single tablet containing magnesium and alpha-lipoic acid supplement or placebo until delivery.

ELIGIBILITY:
Inclusion Criteria:

* 14-34 weeks of gestation

Exclusion Criteria:

* Preexisting diabetes mellitus
* Systolic blood pressure >140mm Hg
* Cancer
* lupus
* hepatitis
* HIV/AIDS
* Diagnosed alcohol or chemical dependency

Ages: 23 Years to 41 Years | Sex: Female
Age Groups: Adult
Dates: Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Number of women with sporadic episodes of preterm uterine contraction | From baseline (beginning of the treatment) until delivery
Number of women with frequent and persistent episodes of preterm uterine contractions associated with pain | From baseline (beginning of the treatment) until delivery
Number of women needed for hospital admission for threatened preterm labour | From baseline (beginning of the treatment) until delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Villa delle Querce, Naples, Italy